**Document Type:** Informed Consent Form

Official Title: National Survey of Young Adult Nutrition (NAYAN)

NCT Number: NCT06096636

**IRB Approval Date:** 06/06/2024

#### CONSENT TO PARTICIPATE IN RESEARCH



**Project Title:** National Survey of Young Adult Nutrition (NAYAN)

Principal Investigators: Julie Hess, Ph.D.; Beth Racine, Ph.D.

Email Addresses: julie.hess@usda.gov; beth.racine@ag.tamu.edu

#### What should I know about this research?

- Taking part in this research is voluntary. Whether you take part is up to you.
- If you don't take part, it won't be held against you.
- You can take part now and later drop out, and it won't be held against you.
- If you don't understand, ask questions. You may contact the researchers above with questions before you consent to the study.
- Ask all the questions you want before you decide.

### How long will I be in this research?

We expect that your taking part in this research will last about one and a half (1.5) hours. You will be asked to answer around 150 questions (30 minutes) and complete a diary of the food and drink you consumed for the prior day (60 minutes). The exact number of questions you answer will depend on your responses, as some questions may have follow-up questions based on how you respond.

### Why is this research being done?

The purpose of this research is to better understand how people's background, habits, and other factors influence their diets and health. We will use this information to help Americans maintain more nutritious diets and improve health.

What happens to me if I agree to take part in this research?

| Approval Date: _ | 6/6/2024 |
|--------------------------------|-----------|
| Expiration Date: | 7/26/2026 |
| University of North Dakota IRB | |

If you decide to take part in this research study, you will fill out a series of questionnaires. These questions will be about you: your demographic information, your beliefs, your attitudes, your knowledge, and your practices.

Some of these questions will be personal. If you feel uncomfortable answering any of these questions, you are free to skip them.

# Could being in this research hurt me?

The risks or discomforts that you may experience from taking part in this research include psychological and/or emotional discomfort because of being asked personal questions.

Additionally, because this research is conducted online, there is always the possibility of a security breach. Given that surveys can be completed from any computer (e.g., personal, work, school), we are unable to guarantee the security of the computer on which you choose to enter your responses. As a participant in our study, we want you to be aware that certain 'key logging' software programs exist that can be used to track or capture data that you enter and/or websites that you visit. To minimize your risk, we recommend that you complete this survey on a private device connected to a private, secure network. Although every reasonable effort has been taken, confidentiality during actual Internet communication procedures cannot be guaranteed.

# Will being in this research benefit me?

It is not expected that you will personally benefit from this research, though you may also gain personal insights because of answering these questions. Possible benefits to others include increased knowledge and understanding of how to improve diets and health.

### How many people will participate in this research?

We expect 1300 people will complete this study conducted by Texas A&M University.

# Will it cost me money to take part in this research?

You will not have any costs for being in this research study. However, you must have access to the Internet. You also need a desktop or laptop computer, smartphone, or tablet on which to complete all the tasks required by this study. Also, we do not withhold income, social security, unemployment taxes, or any other taxes. You may have to pay income taxes on the compensation you receive. All tax questions relating to the taxability of the payment should be directed to your personal tax accountant or to your local Internal Revenue Service Office.

# Will I be paid for taking part in this research?

You will be paid for being in this research study. After completing the questionnaire, you will receive compensation in the amount you have agreed to with the platform through which you entered this survey. After completing the food diary, you will receive a \$35 Amazon gift card code delivered to the email address that you provide on the platform through which you entered this survey.

To protect the integrity of our research, each person is limited to one completion of this survey. If you attempt this survey more than once, you will not receive payment for additional completions. Researchers will review responses to ensure they come from unique individuals.

| Approval Date:6/6/2024 |
|--------------------------------|
| Expiration Date: 7/26/2026 |
| University of North Dakota IRB |

Furthermore, it is important that you read the survey questions and respond truthfully. Researchers will review responses for suspicious activity. If a survey response is flagged for bad responses (for example, clicking through rather than providing genuine responses), you will not receive payment. Participants spending less than 8 minutes (480 seconds) on the questionnaire will not receive payment.

Please note: While you are welcome to skip questions that make you uncomfortable, to receive payment for this survey, you will need to complete at least 90% of the questionnaire and 100% of the dietary recall. If you have skipped less than 10% of the questionnaire and completed the dietary recall, you can expect to receive payment. If you skipped 10% or more of the questionnaire and/or did not complete 100% of the dietary recall, you would not receive payment. If you have concerns regarding the number of questions you skipped, please contact Julie Hess (julie.hess@usda.gov).

There are five questions in the survey that will check for your attention. These questions will have only one correct response. You will be told what the correct response is and instructed to select that correct response. In order to receive payment, you must answer 80% or more of these questions correctly, or at least 4 out of 5 questions. If you answer 3 or fewer of these questions correctly, you will not receive payment.

### Who is funding this research?

This research is being funded by the Texas A&M University Institute for Advancing Health through Agriculture. No one on the research team will receive a direct payment or an increase in salary for conducting this study.

# What happens to information collected for this research?

Your private information may be shared with individuals and organizations that conduct or watch over this research, including:

- The researchers
- People who work with the researchers (support staff)
- The United States Department of Agriculture Agricultural Research Service, as specified in the USDA/ARS Privacy Act System of Records
- The Institutional Review Board (IRB) that reviewed this research

We may publish the results of this research. However, we will keep any identifying information confidential. We protect your information from disclosure to others to the extent required by law. We cannot promise complete secrecy.

Data collected in this research might be de-identified and used for future research or distributed to another investigator for future research without your consent.

#### What if I agree to be in the research and then change my mind?

If you decide to leave the study early, we ask that you send an email to julie.hess@usda.gov to notify us of your withdrawal. You may stop the survey at any time. Your decision will not affect your current or future relations with Texas A&M University.

| Approval Date: _ | 6/6/2024 |
|--------------------------------|-----------|
| Expiration Date: | 7/26/2026 |
| University of North Dakota IRB | |

## Who can answer my questions about this research?

If you have questions, concerns, or complaints, or think this research has hurt you or made you sick, talk to the research team at the email address listed above on the first page.

This research is being overseen by an Institutional Review Board ("IRB"). An IRB is a group of people who perform independent review of research studies. You may talk to them at 701.777.4279 or UND.irb@UND.edu if:

- You have questions, concerns, or complaints that are not being answered by the research team
- You are not getting answers from the research team.
- You cannot reach the research team.
- You want to talk to someone else about the research.
- You have questions about your rights as a research subject.
- You may also visit the UND IRB website for more information about being a research subject: <a href="http://und.edu/research/resources/human-subjects/research-participants.html">http://und.edu/research/resources/human-subjects/research-participants.html</a>

Selecting this box documents your consent to take part in this study.

By selecting this box, I certify that:

- I am 18 years old or older.
- I am a U.S. citizen.
- I have read and agree to the terms above.
- I freely consent to participate in this study.

| $\square$ I am at least 18 years old, a U.S. | citizen, I have read ar | nd agree to the terms | s above, and I freely |
|---|---|---|---|
| consent to participate in this study. | | | |

| Approval Date:6/6/2 | 024 |
|--------------------------------|-------|
| Expiration Date: _7/26/ | /2026 |
| University of North Dakota IRB | |